CLINICAL TRIAL: NCT06714721
Title: Effect of Repetitive Peripheral Magnetic Stimulation on Diaphragm Muscle Thickness, Symptoms and Functional Capacity in Chronic Obstructive Pulmonary Disease
Brief Title: Magnetic Stimulation of Diaphragm in Chronic Obstructive Pulmonary Disease
Acronym: COPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Yeşim Kurtaiş Aytür, MD, Professor, MD, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AU_TTU-2023-3000
Record Dates: First submitted 2024-11-11; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic Obstructive Pulmonary Disease; Pulmonary Rehabilitation; Diaphragm; Repetitive Peripheral Magnetic Stimulation; Strengthening Exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Prospective, sham-controlled, single-blind, randomized controlled trial
Who Masked: Participant
Masking Description: The patients included in the study will be randomized using the Random Allocation Software (RAS) on the computer and divided into two groups: the treatment group and the sham group. All patients will receive an outpatient pulmonary rehabilitation program that includes bronchial hygiene techniques, controlled breathing techniques, respiratory muscle training, aerobic exercises, muscle strengthening, flexibility and stretching, and posture exercises. In addition to the PR program, rPMS will be applied to the patients in the treatment group to stimulate and strengthen the diaphragm muscle. rPMS will be applied to the patients in the sham group without switching it on and a recorded sound of the machine will be played in the background.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group receiving pulmonary rehabilitation and repetitive peripheral magnetic stimulation (Experimental): The treatment group will receive 24 sessions of pulmonary rehabilitation and repetitive peripheral magnetic stimulation to strengthen the diaphragm muscle.
  Interventions: Device: Repetitive peripheral magnetic stimulation
- Sham group (Sham Comparator): The sham group will receive 24 sessions of pulmonary rehabilitation and sham application of repetitive peripheral magnetic stimulation will be done.
  Interventions: Other: Sham (No Treatment)

INTERVENTIONS:
Device: Repetitive peripheral magnetic stimulation — Repetitive peripheral magnetic stimulation treatment will be performed with the "BTL-6000 Super Inductive System Elite" available in our clinic. rPMS treatment will be adjusted to use the stimulus intensity above the motor threshold determined specifically for each patient by selecting the respiratory muscle strengthening protocol set in the device menu. The patient will be given a side-lying position, with the arms in front of the body and the elbows flexed, and the hips and knees in semiflexion. The applicator will be aligned to the diaphragm placement determined by ultrasonography (ninth intercostal space) and placed as close as possible to the skin, and rPMS will be applied for a total of 16 minutes, 8 minutes to the right diaphragm muscle and 8 minutes to the left diaphragm muscle. The treatment period is a total of 16 sessions according to the respiratory muscle strengthening protocol created by the company that developed the device.
  Other Names: BTL-6000 Super Inductive System Elite; rPMS
  Arms: Treatment group receiving pulmonary rehabilitation and repetitive peripheral magnetic stimulation
Other: Sham (No Treatment) — rPMS will be applied to the sham group as sham and the device will not be operated, the applicator of the device will be positioned on the right and left diaphragm muscle for a total of 16 minutes in the same way as the patients in the treatment group, and the sounds recorded during the operation of the device will be played to the patients as if the device was operating in the background. The patients will not know which group they are in.
  Other Names: Sham rPMS
  Arms: Sham group

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a preventable and treatable disease characterized by persistent airflow limitation and respiratory symptoms due to airway and/or alveolar deterioration caused by severe exposure to harmful particles or gases and host factors. Exercise intolerance and decreased functional capacity develop as a result of the disorders that occur in COPD.

The aim of this study is to evaluate the effectiveness of repetitive peripheral magnetic stimulation (rPMS), an easy and inexpensive method to increase diaphragm strength as an adjunct to the pulmonary rehabilitation (PR) program applied in COPD, and to investigate the effect of this method on exercise capacity, diaphragm muscle thickness and symptoms.

DETAILED DESCRIPTION:
COPD is a life-threatening public health problem that starts with shortness of breath, continues with exacerbations, and the prognosis gradually worsens. In COPD patients, respiratory functions decrease due to changes in the airways in the advanced stages of the disease; dyspnea, cough, and sputum emerge as three important symptoms. Respiratory function limitations and symptoms caused by the disease also cause physical and psychological disorders such as peripheral muscle weakness, exercise intolerance, decreased quality of life, depression, and anxiety in patients. Diaphragm dysfunction also develops in COPD. In severe COPD, changes occur in the sarcomere length, enzyme activity, and mitochondrial density of diaphragm muscle fibers. Recurrent COPD attacks also negatively affect diaphragm dysfunction. Due to diaphragm dysfunction, patients' exercise tolerance and daily living activities decrease even more after attacks; their quality of life decreases. The aim of treatment and care in COPD is to prevent progression, reduce symptoms, prevent and/or treat recurrent acute attacks, protect respiratory functions in the long term and prevent functional decline, increase exercise capacity, reduce complications and protect and increase quality of life. Since drug therapy alone is insufficient to achieve these goals, rehabilitation practices should also be a part of the treatment in addition to drug therapy.

Oxygen therapy, nutritional support, pulmonary rehabilitation (PR) approaches are also among the supportive and palliative treatment methods. In the last twenty years, the negative effects of systemic symptoms on the functions of patients in COPD patients have accelerated the development and use of PR. The main goals of PR are to reduce symptoms, bring the person's functional and emotional status to the best possible level, increase participation in daily life and quality of life, and reduce health-related expenses by reversing or stabilizing the systemic effects of the disease. PR has been shown to be the most effective non-pharmacological intervention to improve health status in COPD patients. The main component of PR programs is exercise; which includes aerobic exercise, strengthening exercises, inspiratory muscle training, controlled breathing techniques, bronchial hygiene techniques, stretching exercises, relaxation exercises, as well as water exercises, pilates and yoga programs. There are also daily life activity practices and assistive device training exercises.

Considering the weakness of peripheral muscle and diaphragm muscle strength in COPD patients, alternative strengthening methods for these muscles are important. rPMS is a physical therapy method based on the interaction between a high-intensity electromagnetic field and the human body. The electromagnetic field is generated by a coil placed in the applicator. Depending on the frequency of stimulation and the intensity of the electromagnetic field, it has analgesic, muscle relaxant or muscle strengthening effects. The rPMS method, which is one of the alternative treatment methods that strengthens the diaphragm, does not require direct contact with the skin. Since it can be applied over clothes, the patient does not need to undress or prepare the skin. It is not painful like other invasive methods, so the patient's compliance will be higher and the possibility of abandoning the treatment is less. The rPMS application is fast and easy to use, because there is no need to connect a stimulating electrode to the patient.

In this study, it is planned to investigate the hypothesis that adding rPMS of the diaphragm to the PR program in individuals with COPD would lead to more improvement in exercise capacity, diaphragm muscle thickness, and consequently, symptoms.

In line with this hypothesis, the aim of the study was to evaluate the effectiveness of repetitive peripheral magnetic stimulation (rPMS) to increase diaphragm strength in addition to the PR program applied in COPD, and to investigate the effect of this method on exercise capacity, diaphragm muscle thickness and symptoms.

This is a prospective, randomized, sham-controlled, single-blind, experimental study. Patients who admitt to Ankara University Medical Faculty Hospital Physical Medicine and Rehabilitation Clinic for PR and have stable COPD diagnosis will be invited to the study. This study will be conducted within the scope of good clinical practices and written informed consent forms will be obtained from all patients. The sociodemographic information, smoking history, duration of COPD, presence of co-morbidities, regularly used medications, and other medical history of the patients will be recorded. Patients will be randomized into two groups. Both groups will receive 24 sessions of standard PR programs. Intervention group will also receive repetitive peripheral magnetic stimulation (rPMS) to strengthen the diaphragm muscle. Patients will be evaluated at baseline and at the end of the program. The assessments will include cardiopulmonary exercise test (CPET) for dynamic respiratory functions and VO2max and six-minute walk test to determine functional exercise capacity, Saint George Respiratory Questionnaire (SGRQ) for health specific quality of life, Transitional Dyspnea Index (TDI) measuring changes in shortness of breath, Modified Medical Research Council (mMRC) Dyspnea Scale and diaphragm muscle thickness measurement with ultrasonography.

ELIGIBILITY:
Inclusion Criteria:

1. Having been diagnosed with COPD at least 6 months ago
2. Being over 18 years of age
3. Having the cognitive ability to understand the questions and fill out the questionnaires
4. Agreeing to participate in the study

Exclusion Criteria:

1. Presence of chest wall deformity
2. Presence of pacemaker/defibrillator
3. Pregnancy
4. Presence of acute respiratory tract infection and/or pneumonia
5. Suspicion of underlying hemidiaphragmatic paresis (defined as elevation of one hemidiaphragm >2.5 cm compared to the other on chest radiography)
6. Known history of inflammatory rheumatologic or neuromuscular disease that may affect the mechanics of the diaphragm (cerebrovascular accident, spinal cord injury, epilepsy, peripheral neuropathy, and muscle diseases, etc.)
7. Suspected paraneoplastic or myopathic syndromes and/or use of medications known to alter muscle structure and/or function, including oral corticosteroids
8. History of recent thoracic and/or abdominal surgery
9. History of COPD exacerbation within the last 4 weeks
10. COPD disease is accompanied by bronchial asthma, interstitial lung diseases, lung neoplasia, metabolic diseases (diabetes mellitus, uremia and liver failure)
11. Body mass index greater than 40
12. Presence of contraindications for exercise program (uncontrolled atrial/ventricular arrhythmia, resting systolic blood pressure ≥ 200 mm Hg or diastolic blood pressure ≥ 110 mm Hg, severe aortic stenosis, recent history of embolism, decompensated heart failure, cardiac ischemic event within the last four weeks)
13. Presence of systemic disease and/or musculoskeletal disease that may prevent exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-08-23 (Actual); Primary Completion 2025-08-04 (Estimated); Study Completion 2025-12-04 (Estimated)

PRIMARY OUTCOMES:
Maximum oxygen consumption (VO2max) | From enrollment to the end of treatment at 6 weeks
  V̇O2 max (also maximal oxygen consumption, maximal oxygen uptake or maximal aerobic capacity) is the maximum rate of oxygen consumption attainable during physical exertion. It reflects cardiorespiratory fitness and endurance capacity in exercise performance and is accepted as the gold standard for the maximal exercise capacity of an individual. As part of the study, patients will undergo cardiopulmonary exercise testing (CPET) twice, before and after treatment.The cardiopulmonary exercise test will be applied on the treadmill under the supervision of a doctor and a physiotherapist. The aim of the test is to measure the maximum oxygen consumption of the patients (VO2max); therefore, the test protocol appropriate to the patient's current condition will be selected.

SECONDARY OUTCOMES:
6-minute walk test (6MWT) | From enrollment to the end of treatment at 6 weeks
  The 6-minute walk test is used to measure functional capacity in people with lung disease, to evaluate medical practices, response to pulmonary rehabilitation, course of disease, and to assess disability caused by pulmonary problems. It allows for accurate calculation of exercise tolerance and functional capacity. Healthy individuals can walk distances of 400-700 m in six minutes. The 6-minute walk test will be performed in the 30-meter test corridor. Before starting the test, patients will be asked to rest for at least 10 minutes. Patients will be asked to walk in the corridor as fast as they can for 6 minutes. The total distance they have walked will be determined . Heart rate, blood pressure, and oxygen saturation will be COPD has been shown to be associated with increased mortality with a six-minute walk distance of < 350 m. An increase of 30 m (25-33 m) in the 6-minute walk test is considered to reflect clinically significant improvement.
Diaphragm thickness measurement | From enrollment to the end of treatment at 6 weeks
  Diaphragm thickness will be measured by ultrasonographic evaluation. It will be performed using a linear array transducer (7-12 MHz) with an ultrasound scanner (LogiqP5, GE Medical Systems). Measurements will be made with the patient in the supine position. The diaphragm will be imaged by placing the transducer in the ninth intercostal space between the patient's anterior and midaxillary lines, perpendicular to the two ribs. Diaphragm thickness measurements will be made at the end of expiration. The average value of three consecutive measurements will be recorded.
Health-related quality of life | From enrollment to the end of treatment at 6 weeks
  St. George Respiratory Questionnaire (SGRQ) is specific for respiratory diseases measuring health-related quality of life. SGRQ questions 50 items divided into three domains: symptoms (8 items), activities (16 items), effects of the disease (26 items). Symptoms domain questions the patient's respiratory discomfort and the level of cough, sputum, wheezing in the chest and shortness of breath. The activity component is related to physical activities that can cause shortness of breath or are restricted due to shortness of breath. The impact component covers factors such as work, occupation, keeping one's health under control, panic, medication and its side effects, and discomfort during daily life activities. The three sections of the test are scored separately and the total score is calculated. Scores range from 0 to 100, zero indicating normal and 100 indicating severe limitation. A change of four units for the total score and/or each subsection is accepted clinically significant.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University Faculty of Medicine Department of Physical Medicine and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared when asked for systemic or meta analyses.